CLINICAL TRIAL: NCT03832075
Title: Validity of Korebalance Balance System in Postmenopausal Osteoporotic Patients
Brief Title: Validity of Korebalance Balance System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Bilinç Doğruöz Karatekin, MD, Research Assistant of PMR, Istanbul Medeniyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MedeniyetOP2
Record Dates: First submitted 2019-02-02; First posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Osteoporosis, Postmenopausal; Balance; Distorted
Keywords: osteoporosis; balance; berg balance scale; korebalance balance system
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- postmenopausal osteoporosis (Experimental): Postmenopausal osteoporotic patients evaluated with Berg Balance Scale, Timed Up and Go test and Korebalance balance system for balance disorder.
  Interventions: Diagnostic Test: Berg Balance Scale; Diagnostic Test: Timed Up and Go Test; Diagnostic Test: Korebalance Balance System

INTERVENTIONS:
Diagnostic Test: Berg Balance Scale — Berg Balance Scale is 14 item scale for detecting balance disorder.
Diagnostic Test: Timed Up and Go Test — Timed Up and Go Test assesses mobility, balance, walking ability, and fall risk in older adults.
Diagnostic Test: Korebalance Balance System — Korebalance Balance System evaluates the balance and stability using objective neuro-sensory balance assessment. Static Test requires standing steady & balancing on the platform, keeping the crosshairs of cursor in the center of the test pattern. The Score indicates the deviation of user's center of gravity from the center of the pattern. Dynamic Test offers a moving cursor that the user "follows". Four patterns are offered: Circle, Square, Infinity and Random. Each pattern is available in three dimensions: Small, Medium and Large; five speeds; Clockwise and Counterclockwise directions.

SUMMARY:
In postmenopausal osteoporosis patients, the balance is impaired. Equilibrium is evaluated with various test and balance systems. This study aims evaluation of the patients with the Korebalance Balance System and balance tests and investigation the validity of the Korebalance Balance System.

DETAILED DESCRIPTION:
53 postmenopausal osteoporosis patients were evaluated with balance tests (Berg Balance Scale (BBS) and Timed Up and Go Test (TUG)) and Korebalance Balance System. The Korebalance Balance System is a balance assessment and exercise system. The higher the score, the greater the deterioration in the balance. The results of static and dynamic balance evaluation are recorded as score values. In this study, investigators compared Korebalance Balance System, Berg Balance Scale (BBS) and Timed Up and Go (TUG) tests and other demographic and clinical parameters (age, body mass index (BMI), 25OHvitD level, menopause age, fall within the last 1 year, fracture history, history of fracture in mother).

ELIGIBILITY:
Inclusion Criteria:

* Having postmenopausal osteoporosis
* No other disease that can cause balance disorder
* Volunteer participation in the study

Exclusion Criteria:

* To have a disease that will cause balance disorder,
* Having understanding problem to prevent communication with the patient,
* The lack of motor function to the balance device.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal osteoporotic patients
Enrollment: 53 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Evaluate validity of Korebalance Balance System in postmenopausal osteoporotic patients | 6 months
  The statistical correlation of Korebalance Balance System and Berg Balance Scale was investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University Faculty of Medicine, Physical Therapy and Rehabilitation Department, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided